CLINICAL TRIAL: NCT06627816
Title: Efficacy of Intravenous Nefopam, Dexmedetomidine, and Meperidine in Preventing Post-Spinal Anesthesia Shivering in Adult Patients Undergoing Lower Abdominal and Lower Limb Surgeries: A Double-Blind Comparative Study
Brief Title: Efficacy of Intravenous Nefopam, Dexmedetomidine, and Meperidine in Preventing Post-Spinal Anesthesia Shivering in Adult Patients Undergoing Lower Abdominal and Lower Limb Surgeries.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Amany Ahmed Eissa, lecturer of anesthesia& ICU, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: N-343-2024
Record Dates: First submitted 2024-10-03; First posted 2024-10-04 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Nefopam; Dexmeditomidine; Meperidine; Post-spinal Anesthesia Shivering
MeSH Terms: interventions — Nefopam; Meperidine

STUDY DESIGN:
Intervention Model Description: comparative study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- nefopam group (Active Comparator): • Group N (n=80) will receive nefopam 0.15 mg/kg i.v. (Nopain®, Medical Union Pharmaceuticals MUP, Ismailia, Egypt, Ampoules of 20 mg/1 ml)
  Interventions: Drug: Nefopam
- dexmeditomidine group (Active Comparator): • Group D (n=80) will receive dexmedetomidine 0.5 µg/kg i.v. (Precedex®, Hospira Inc, USA, Vials of 200 mg/2 ml)
  Interventions: Drug: Nefopam
- meperidine group (Active Comparator): • Group P (n =80) will receive pethidine (meperidine) 0.5 mg/kg i.v. (Ampoules of 50 mg/1 ml).
  Interventions: Drug: Nefopam

INTERVENTIONS:
Drug: Nefopam — efficacy of 3 drugs in preventing post-spinal anesthesia shivering
  Other Names: dexmeditomidine; meperidine

SUMMARY:
This prospective, randomized, controlled, double-blinded study is designed to evaluate the efficacy of nefopam compared to dexmedetomidine and meperidine for the prevention of postspinal anesthesia shivering while minimizing side effects.

DETAILED DESCRIPTION:
Numerous clinical studies have demonstrated that nefopam effectively prevents and treats postoperative shivering after general anesthesia. For instance, a dose of 0.15 mg/kg nefopam is comparable in efficacy to 0.5 µg/kg dexmedetomidine for treating shivering after orthopedic or abdominal surgery. Additionally, 20 mg of nefopam is equally effective as 50 mg of meperidine in preventing shivering following certain neurosurgical procedures . Notably, patients administered nefopam experience less sedation and hypotension compared to those given dexmedetomidine. However, further research is needed to evaluate nefopam's effects on preventing shivering after neuraxial blockades.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 21-60 undergoing elective lower abdominal, urological, gynecological, lower limb, orthopedic, or plastic surgeries under spinal anesthesia.

  * ASA physical status I and II.

Exclusion Criteria:

* • Known hypersensitivity to nefopam, dexmedetomidine, or pethidine.

  * Thyroid disorders, psychiatric disorders, severe diabetes, or autonomic neuropathies
  * Known history of substance or alcohol abuse
  * A history of convulsive disorders or severe neurological diseases
  * Severe cardiac, pulmonary, renal, or hepatic disease
  * Obstetric procedures and procedures requiring transfusion of blood and blood products.
  * A contraindication to spinal anesthesia, e.g., coagulation disorders, local or general infection, increased intracranial tension, and progressive neurological disorders.
  * Failed or partial spinal block.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-07-05 (Actual)

PRIMARY OUTCOMES:
the incidence of shivering during the whole observation period | 120 minutes
  shivering score ≥ 3. The shivering score will be assessed at 10-minute intervals after the spinal block and graded by the scale validated by Wrench et al.

SECONDARY OUTCOMES:
- Intraoperative hemodynamic variables | 120 minutes
  - (HR, MAP, SPO2) every 15 minutes
axillary body temperature | 120 minutes
  every 30 minutes
recurrent shivering | 120 minutes
  response to treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Al Aini Hospitals, Cairo, Egypt

REFERENCES:
- [Derived] Abdelhafez EM, El-Siory W, Turki D, Eissa AA. Efficacy of Intravenous Nefopam, Dexmedetomidine, and Meperidine in Preventing Postspinal Anesthesia Shivering in Adult Patients Undergoing Lower Abdominal and Lower Limb Surgeries: A Double-Blind Comparative Study. Anesthesiol Res Pract. 2025 Dec 3;2025:4549345. doi: 10.1155/anrp/4549345. eCollection 2025. PMID 41346412